CLINICAL TRIAL: NCT04623333
Title: A Single-arm, Open-label, Multicenter, Phase II Study of TQB2450 Injection in Subjects With PD-L1 Positive Recurrent or Metastatic Cervical Cancer
Brief Title: A Study of TQB2450 Injection in Subjects With PD-L1 Positive Recurrent or Metastatic Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-II-09
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-08

CONDITIONS: Recurrent or Metastatic Cervical Cancer
MeSH Terms: conditions — Recurrence; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450 injection (Experimental): TQB2450 1200mg administered intravenously (IV) on Day 1 of each 21-day cycle.
  Interventions: Drug: TQB2450

INTERVENTIONS:
Drug: TQB2450 — TQB2450 1200mg administered intravenously (IV) on Day 1 of each 21-day cycle.

SUMMARY:
This is a study to evaluate the efficacy and safety of TQB2450 injection in the treatment of PD-L1 positive recurrent or metastatic cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understood and signed an informed consent form; 2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months; 3. Diagnosed as recurrent or metastatic cervical cancer; 4. Has received ≥first-line platinum-containing chemotherapy, and disease progress or recur during or after treatment; 5. PD-L1 positive, and the combined positive score (CPS) ≥1; 6. Has at least one measurable lesion; 7. Adequate laboratory indicators; 8. Serum or urine pregnancy tests are negative within 7 days before randomization; Men and women should agree to use effective contraception during the study period and after the end of the study period within 6 months.

Exclusion Criteria:

* 1. Combined diseases and medical history: a) Has diagnosed and/or treated additional malignancy within 3 years prior to first dose;b) Diagnosed as other special pathological types, such as mucinous adenocarcinoma, clear cell adenocarcinoma, neuroendocrine tumor and so on;c) Unalleviated toxicity ≥ grade 1 due to any previous anticancer therapy;d) Has received major surgical treatment, open biopsy and so on within 28 days before the start of the study;e) Has a unhealed wound or fracture for a long time; f) Has cerebrovascular accident, deep vein thrombosis and pulmonary embolism within 6 months before the study; g) Has a history of psychotropic substance abuse and unable to quit or mental disorders; h)Has any serious and / or uncontrolled disease; 2.Tumor-related symptoms and treatment: a) Has received surgery, chemotherapy, radiotherapy or other anticancer therapy within 4 weeks before the start of the study; b) Has received proprietary Chinese medicine with anti-tumor indications in the NMPA approved drug instructions within 2 weeks before the start of the study; c) Has received immunotherapeutic drugs against PD-1, PD-L1, CTLA-4 and other related drugs; d) Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage; e) Has symptomatic central nervous system (CNS) disease and/or cancerous meningitis, pia mater disease; 3. Related to treatment of research: a) Has received attenuated live vaccine within 28 days before first dose or planned to received attenuated live vaccine during the study period; b) Has severe hypersensitivity reactions after using monoclonal antibodies; c) Has active autoimmune diseases requiring systemic treatment occurred within 2 years before the study; d) Has a history of active tuberculosis; 4.Has Participated in other clinical trials within 4 weeks before first dose. 5.According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) evaluated by Independent Review Committee (IRC) | up to 12 months
  ORR defined as percentage of participants achieving complete response (CR) and partial response (PR), recorded from the first dose until the first documented progressive disease (PD) or death from any cause, based on IRC.

SECONDARY OUTCOMES:
Overall response rate (ORR) evaluated by investigator | up to 12 months
  ORR defined as percentage of participants achieving complete response (CR) and partial response (PR), recorded from the first dose until the first documented progressive disease (PD) or death from any cause, based on investigator.
Disease Control Rate (DCR) | up to 12 months
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of response (DOR) | up to 12 months
  The time when the participants first achieved complete or partial remission to disease progression.
Progression free survival (PFS) | up to 12 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | up to 18 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
DOR rate (≥ 6 months) | up to 12 months
  The percentage of participants achieved complete or partial remission ≥ 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shangdong, China